CLINICAL TRIAL: NCT06814964
Title: A Phase I Pilot Clinical Trial of Dose Escalation With Stereotactic-Guided Intraventricular Thrombolysis Using Tenecteplase (rhTNK-tPA) for Intraventricular Hemorrhage.
Brief Title: rhTNK-tPA Thrombolytic Removal of Intraventricular Hemorrhage
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Dr. Yong Cao, Chief Physician, Beijing Tiantan Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: rhTNK-tPA-IVH01
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-01

CONDITIONS: Intraventricular Hemorrhage
Keywords: intraventricular hemorrhage; Stereotactic puncture therapy; rhTNK-tPA
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low dose rhTNK-tPA thrombolytic removal of intraventricular hemorrhage (Experimental): Low dose tenecteplase (injection amount = volume of intraventricular hematoma × 0.009 mg/ml) was diluted to 1ml with sterile injection water, and administered via the EVD. At least 4 ml of CSF is removed prior to injection of 1 ml of test article followed by a 3 ml flush of sterile saline into the ventricle. Injection is followed by closure of the catheter for 1 hour and then opening of the EVD for drainage of clot and CSF until the next injection every 12 hours. Treatment continues for up to 8 doses of test article unless, an treatment success endpoint of clot lysis is reached, or an adverse treatment endpoint occurs (e.g. new hemorrhage: compared with the previous time point CT, a CT value of > 72Hu and a volume of > 5ml). Treatment success endpoints are (i) both 3rd and 4th ventricles are open; (ii) IVH related mass effect [dilated or shifted ventricle] is resolved; or (iii) an estimated 80% resolution of the IVH clot has occurred from the time clot stability was established.
  Interventions: Drug: Low dose group
- Medium dose rhTNK-tPA thrombolytic removal of intraventricular hemorrhage (Experimental): Medium dose tenecteplase (injection amount = volume of intraventricular hematoma × 0.018 mg/ml) was diluted to 1ml with sterile injection water, and administered via the EVD. At least 4 ml of CSF is removed prior to injection of 1 ml of test article followed by a 3 ml flush of sterile saline into the ventricle. Injection is followed by closure of the catheter for 1 hour and then opening of the EVD for drainage of clot and CSF until the next injection every 12 hours. Treatment continues for up to 8 doses of test article unless, an treatment success endpoint of clot lysis is reached, or an adverse treatment endpoint occurs (e.g. new hemorrhage: compared with the previous time point CT, a CT value of > 72Hu and a volume of > 5ml). Treatment success endpoints are (i) both 3rd and 4th ventricles are open; (ii) IVH related mass effect [dilated or shifted ventricle] is resolved; or (iii) an estimated 80% resolution of the IVH clot has occurred from the time clot stability was established.
  Interventions: Drug: Medium dose group
- High dose rhTNK-tPA thrombolytic removal of intraventricular hemorrhage (Experimental): High dose tenecteplase (injection amount = volume of intraventricular hematoma × 0.027 mg/ml) was diluted to 1ml with sterile injection water, and administered via the EVD. At least 4 ml of CSF is removed prior to injection of 1 ml of test article followed by a 3 ml flush of sterile saline into the ventricle. Injection is followed by closure of the catheter for 1 hour and then opening of the EVD for drainage of clot and CSF until the next injection every 12 hours. Treatment continues for up to 8 doses of test article unless, an treatment success endpoint of clot lysis is reached, or an adverse treatment endpoint occurs (e.g. new hemorrhage: compared with the previous time point CT, a CT value of > 72Hu and a volume of > 5ml). Treatment success endpoints are (i) both 3rd and 4th ventricles are open; (ii) IVH related mass effect [dilated or shifted ventricle] is resolved; or (iii) an estimated 80% resolution of the IVH clot has occurred from the time clot stability was established.
  Interventions: Drug: High dose group

INTERVENTIONS:
Drug: Low dose group — The calculated injection amount of tenecteplase (tenecteplase injection amount = volume of intraventricular hematoma × 0.009 mg/ml) was diluted to 1ml with sterile injection water, and administered via the EVD.
  Arms: Low dose rhTNK-tPA thrombolytic removal of intraventricular hemorrhage
Drug: Medium dose group — The calculated injection amount of tenecteplase (tenecteplase injection amount = volume of intraventricular hematoma × 0.018 mg/ml) was diluted to 1ml with sterile injection water, and administered via the EVD.
  Arms: Medium dose rhTNK-tPA thrombolytic removal of intraventricular hemorrhage
Drug: High dose group — The calculated injection amount of tenecteplase (tenecteplase injection amount = volume of intraventricular hematoma × 0.027 mg/ml) was diluted to 1ml with sterile injection water, and administered via the EVD.
  Arms: High dose rhTNK-tPA thrombolytic removal of intraventricular hemorrhage

SUMMARY:
The purpose of this pilot study is to determine the safety and optimal dose of clot lysis with rhTNK-tPA for intraventricular hemorrhage, using stereotactic guidance for extraventricular drain placement.

DETAILED DESCRIPTION:
In patients with spontaneous intracerebral hemorrhage (ICH), intraventricular hemorrhage (IVH) is often associated with catastrophic outcomes. Studies have reported that the mortality rate in ICH patients with IVH exceeds 50%, and fewer than 20% of survivors achieve good functional outcomes. Hematoma lysis therapy appears to influence both mortality and functional recovery. Previous systematic reviews and meta-analyses suggest that the removal of intraventricular hemorrhage, by alleviating acute obstructive hydrocephalus and reducing neurotoxicity, may improve survival rates and long-term functional outcomes. The CLEAR III trial, published in The Lancet, demonstrated that in patients with IVH and external ventricular drainage, the 180-day mortality rate was lower with intraventricular alteplase lavage compared to saline (0.9%), although functional outcomes did not improve.

Alteplase, a second-generation fibrinolytic agent, facilitates the dissolution of hematomas following intraventricular hemorrhage. However, its low fibrin specificity, short half-life, and weak resistance to plasminogen activator inhibitor type 1 (PAI-1) often necessitate multiple thrombolytic administrations. This may explain the lack of improvement in neurological functional outcomes. In contrast, tenecteplase, a third-generation fibrinolytic agent, exhibits higher fibrin specificity and a longer half-life, which may enhance thrombolytic efficiency and hematoma clearance rates. These properties make tenecteplase a potentially safer and more effective option for hematoma dissolution in patients with intraventricular hemorrhage.

Building on the findings of the CLEAR III trial and previous research, this study aims to replace alteplase with tenecteplase and conduct a prospective, single-center, "3+3" dose-escalation trial to evaluate the safety and optimal dosing of tenecteplase-assisted hematoma dissolution for intraventricular hemorrhage. The results will provide a foundation for future multicenter randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years.
2. Symptom onset within 24 hours prior to diagnostic CT scan. Patients with unknown onset time should be excluded. For patients with symptoms occurring during sleep, the time of symptom onset should be considered as the last time the patient was awake and asymptomatic.
3. Spontaneous intracerebral hemorrhage (ICH) ≤ 30 ml，with intraventricular hemorrhage (IVH) >20 ml obstructing the third and/or fourth ventricles.
4. All patients must have an external ventricular drain (EVD) placed prior to enrollment: The EVD should be accurately positioned into the largest cerebrospinal fluid (CSF) pool or the least bloody site in the lateral ventricle using robotic stereotactic guidance.
5. A stability CT scan performed ≥ 6 hours after EVD placement must confirm ICH clot stability: The ICH volume change should be ≤ 5 ml compared to the previous CT scan. If the stability CT scan shows a difference > 5 ml, a repeat stability CT scan should be performed ≥ 12 hours later. Stability CT scans may be repeated every 12 hours within 72 hours of the diagnostic CT scan. If two consecutive CT scans show a hematoma enlargement ≤ 5 ml and the ICH volume remains ≤ 35 ml, the patient is eligible.
6. IVH clot stability: The width of the lateral ventricle most affected by the clot must not increase by > 2 mm. If the stability CT scan shows a difference > 2 mm, a repeat stability CT scan should be performed ≥ 12 hours later. Stability CT scans may be repeated every 12 hours within 72 hours of the diagnostic CT scan. If two consecutive CT scans show a change ≤ 2 mm, the patient is eligible.
7. Catheter tract bleeding on the stability CT scan must be ≤ 5 ml. If any CT slice shows catheter tract bleeding > 5 ml, a repeat stability CT scan should be performed ≥ 12 hours later. Stability CT scans may be repeated every 12 hours within 72 hours of the diagnostic CT scan. If two consecutive CT scans show a change ≤ 5 ml and the total hematoma volume along the tract is ≤ 10 ml, the patient is eligible.
8. On the stability CT scan, the third and/or fourth ventricles must be occluded with blood.
9. Primary IVH (ICH = 0) is eligible.
10. Sustained systolic blood pressure (SBP) < 180 mmHg for at least 6 hours prior to enrollment. (Patients do not need to meet the SBP criteria throughout the screening period, but vital signs should remain stable during the enrollment window).
11. No intraventricular thrombolytic treatment within 12 hours of symptom onset.
12. Enrollment must be completed within 72 hours of the diagnostic CT scan. (The 72-hour limit may be extended with PI approval for reasons such as hematoma stability, INR stability, or other valid justifications).
13. Pre-morbid modified Rankin Scale (mRS) score of 0 or 1.

Exclusion Criteria:

1. Hemorrhage caused by aneurysms, arteriovenous malformations (AVM), tumors, or other identifiable causes. If the cause of ICH is unknown, CTA, DSA, or other definitive imaging must be performed during screening to rule out these causes. If imaging is negative, the patient is eligible.
2. Presence of choroid plexus vascular malformation or Moyamoya disease.
3. Hypercoagulable state or coagulopathy. Patients requiring long-term anticoagulation are excluded. Reversal of anticoagulation is permitted if long-term anticoagulation is not required.
4. Use of anticoagulants (e.g., dabigatran, apixaban, rivaroxaban) or antiplatelet agents (e.g., tirofiban, ticagrelor, cilostazol, clopidogrel) within one week prior to symptom onset (aspirin is allowed).
5. Platelet count < 100,000 or INR > 1.4.
6. Pregnancy (positive serum or urine pregnancy test).
7. Infratentorial hemorrhage.
8. Thalamic hemorrhage with significant midbrain extension, third nerve palsy, or dilated and non-reactive pupils. Other supranuclear gaze abnormalities are not excluded. Posterior fossa or cerebellar hemorrhages are excluded.
9. Subarachnoid hemorrhage (SAH) or any atypical hematoma location or appearance on diagnostic CT scan. Angiography (CTA, DSA, or MRA/MRI) must be performed to rule out other causes. If no source of bleeding is identified, the patient is eligible. Cortical SAH secondary to clot lysis is eligible.
10. Unstable ICH/IVH with ongoing hematoma enlargement.
11. Indications for craniotomy: ① Progressive decline in consciousness; ② Signs of brain herniation; ③ Hematoma located < 1 cm from the cortical surface.
12. Ongoing internal bleeding involving retroperitoneal, gastrointestinal, genitourinary, or respiratory tracts. Patients with prior bleeding that is clinically stable for ≥ 12 hours and without coagulopathy or bleeding disorders are eligible.
13. Multifocal superficial bleeding at multiple vascular puncture or access sites (e.g., venipuncture, arterial puncture) or recent surgical sites.
14. Any condition that, in the investigator's opinion, poses a significant risk to the patient or makes the patient unsuitable for the study.
15. Planned or concurrent participation in another interventional clinical trial. Participation in observational, natural history, or epidemiological studies without intervention is allowed.
16. Inability to obtain informed consent from the patient or legal representative.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Drug-related new rebleeding events | 24, 48, 72, and 96 hours after the first dose tenecteplase administration.
  CT examinations were performed every 24 hours after tenecteplase administration. Compared with the CT at the previous time point, a CT value of more than 72 HU and a volume of more than 5 ml were defined as newly emitted blood.

SECONDARY OUTCOMES:
Mortality rate | within 7 days of enrollment
  Death within 7 days of enrollment
Ventricular infection | within 7 days of enrollment
  fever and positive cerebrospinal fluid culture
Clot Removal | 24 hours after the last dose.
  Change in blood volume measured between stability scan and 24 hours after the last dose.
Number of doses administered at the endpoint of the treatment | 24, 48, 72, and 96 hours after the first dose tenecteplase administration.
  Record the number of doses administered at the endpoint of the treatment.
The rate of resolution of 3rd and/or 4th ventricles obstruction at the endpoint of treatment. | 24, 48, 72, and 96 hours after the first dose tenecteplase administration.
  CT examinations were performed every 24 hours after tenecteplase administration to determine the resolution of 3rd and/or 4th ventricles obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Cao, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided